CLINICAL TRIAL: NCT07379138
Title: Launching the Era of Melanoma Survivorship: Defining Benchmarks in Quality of Life Inclusive of Mental Health (QOL-MH)
Brief Title: Studying Quality of Life Inclusive of Mental Health and Cognitive Behavioral Therapy for Cancer Distress for the Improvement of Quality of Life in Stage III-IV Melanoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-007199; NCI-2026-00039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-007199 (Other: Mayo Clinic Institutional Review Board); HT9425-25-1-0802 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Practice Guidelines as Topic; Standard of Care; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 1 (QOL-MH) (Experimental): Patients complete QOL-MH questionnaires at baseline and 3, 6, 9, 12, 18, and 24-months post-stage III-IV diagnosis. Patients living in Minnesota, Iowa, or Wisconsin may also optionally participate in aim 2.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration
- Aim 2 arm I (CBT-C) (Experimental): Patients attend CBT-C sessions once a week for 6 weeks in the absence of unacceptable toxicity.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Aim 2 arm II (SOC) (Active Comparator): Patients receive SOC for 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC
  Other Names: standard of care; standard therapy
  Arms: Aim 2 arm II (SOC)
Behavioral: Cognitive Behavior Therapy — Attend CBT-C sessions
  Other Names: CBT; cognitive therapy; CT
  Arms: Aim 2 arm I (CBT-C)
Other: Electronic Health Record Review — Ancillary studies
Other: Questionnaire Administration — Complete QOL-MH questionnaires

SUMMARY:
This clinical trial studies how people feel and live during the first two years after being treated for melanoma and whether cognitive behavioral therapy for cancer distress (CBT-C) works to improve quality of life in patients with stage III-IV melanoma. The melanoma survivorship population is rapidly growing, given the increasing survival rates due to treatment advancements. An urgent need to better define and optimize comprehensive quality of life inclusive of mental health (QOL-MH) has been identified. Cognitive behavioral therapy is a type of psychotherapy that helps patients change their behavior by changing the way they think and feel about certain things. CBT-C is a new type of care that helps patients cope with cancer-related stress, which can include problems like trouble sleeping, trouble focusing, or changes in social life and daily activities. Gathering information on how melanoma patients feel and live during the first two years after treatment may help promote improved care and continued scientific advancements in the understanding of melanoma specific QOL-MH and survivorship as a whole, and may also help determine whether CBT-C improves qualify of life in patients with stage III-IV melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18-years
* Stage III-IV melanoma and =< 2 month duration of this diagnosis
* Able to read English sufficient to complete survey, informed consent

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in FACT-M total score (Aim 1) | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Functional Assessment of Cancer Therapy - Melanoma (FACT-M) is a 52-item questionnaire used to measures quality of life (QoL) in melanoma cancer patients. Responses to each item are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Scores range from 0-108 with higher scores indicating better quality of life. For this study, 8 items have been omitted, so the number of items is 44, with total scores ranging from 0-176. Descriptive statistics will be used to tabulate and graph the observed total scores and the change from baseline total scores over time.
Change in FACT-ICM total score (Aim 1) | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Functional Assessment of Cancer Therapy - Immune Checkpoint Modulator (FACT-ICM) is a 25-item subscale that measures symptom burden and health-related quality of life (HRQoL) over the past 7 days in patients receiving immune checkpoint inhibitors. Responses to each question are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Scores range from 0-100 with higher scores indicating greater symptom burden and poorer quality of life. Descriptive statistics will be used to tabulate and graph the observed total scores and the change from baseline total scores over time.
Change in Impact of Events Scale-Revised (IES-R) score (Aim 1) | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Impact of Event Scale-Revised (IES-R) is a 22-item self-report measure designed to assess subjective distress related to stressful life events. The IES-R consists of 22 items for which participants rate how distressing each difficulty has been during the past 7 days with regard to their cancer diagnosis. Responses are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Scores range from 0-88 with higher scores indicating greater distress. Descriptive statistics will be used to tabulate and graph the observed total scores and the change from baseline total scores over time.
Change in IES-R score (Aim 2) | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Impact of Event Scale-Revised (IES-R) is a 22-item self-report measure designed to assess distress related to stressful life events. The IES-R consists of 22 items which participants rate distress over the past 7 days with regard to their cancer diagnosis. Responses are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Scores range from 0-88 with higher scores indicating greater distress.

SECONDARY OUTCOMES:
Change in PHQ-8 score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Patient Health Questionnaire-8 (PHQ-8) is a brief, self-report tool used to screen for and measure the severity of depression by asking about 8 depressive symptoms over the past two weeks, scoring from 0 (not at all) to 3 (nearly every day) for each, with total scores indicating severity (e.g., 0-4 minimal, 10-14 moderate) and a score of 10 or more often suggesting major depression.
Change in GAD-7 Anxiety score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The General Anxiety Disorder 7-item (GAD-7) scale is used to assess symptoms and feelings of anxiety over the past two weeks. The GAD-7 consists of 7 questions answered on a scale of 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21 where 0 indicates no anxiety, 1-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. If patients indicate any problems they are asked to indicate how difficult the problems have made daily life: not difficult at all, somewhat difficult, very difficult, or extremely difficult.
Change in PSQI score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Pittsburgh Sleep Quality Index (PSQI)measures the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.
Change in PROMIS: Fatigue score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS): Fatigue questionnaire, a subscale of the PROMIS-29, measures fatigue and related symptoms over the past seven days. It consists of four items rated on a scale of 1(not at all) to 5 (very much). A higher score indicates greater experience of fatigue.
Change in PROMIS: Pain Interference score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The PROMIS: Pain Interference questionnaire, a subscale of the PROMIS-29, is used to assess pain interference in daily life over the past seven days. It consists of four items rated on a scale of 1(not at all) to 5 (very much). A higher score indicates greater levels of pain interference.
Change in COST-FACIT score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COSTFACIT) measures financial toxicity among cancer patients. This measure reflects five themes of financial toxicity which include: financial, resource, affect, coping, and effect on family. It consists of 12 questions, each answered on a scale of 0 (not at all) to 5 (very much), with higher scores indicating greater financial toxicity.
Change in MEPS score | Baseline (at enrollment) and 3, 6, 9, 12, 18, and 24 months
  The Medical Expenditures Survey (MEPS) measures the financial impact of cancer, its treatment, or the lasting effects of that treatment. It consists of 5 multiple choice questions, including free text/ / fill-in options where appropriate. Results are reported descriptively. .

CONTACTS AND LOCATIONS:
Overall Officials: Shawna L. Ehlers, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials